CLINICAL TRIAL: NCT06277284
Title: A Randomized, Open, Parallel, Phase I Clinical Trial Comparing the Pharmacokinetics of MG-K10 Humanized Monoclonal Antibody in Healthy Adults
Brief Title: Clinical Study of MG-K10 Humanized Monoclonal Antibody Injection in Healthy Adult Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Collaborators: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MG-K10-I-002
Record Dates: First submitted 2023-10-23; First posted 2024-02-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-10

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MG-K10 humanized monoclonal antibody injection (prefilled syringe) (Experimental): single injection
  Interventions: Drug: MG-K10 humanized monoclonal antibody injection (prefilled syringe)
- MG-K10 humanized monoclonal antibody injection (Active Comparator): single injection
  Interventions: Drug: MG-K10 humanized monoclonal antibody injection（Penicillin bottle）

INTERVENTIONS:
Drug: MG-K10 humanized monoclonal antibody injection (prefilled syringe) — MG-K10 Humanized Monoclonal Antibody Injection
  Other Names: MG-K10 (prefilled syringe)
  Arms: MG-K10 humanized monoclonal antibody injection (prefilled syringe)
Drug: MG-K10 humanized monoclonal antibody injection（Penicillin bottle） — MG-K10 humanized monoclonal antibody injection (single injection)
  Other Names: MG-K10 （Penicillin bottle）
  Arms: MG-K10 humanized monoclonal antibody injection

SUMMARY:
Research Topics A randomized, open-label, parallel-group, phase I clinical trial comparing the pharmacokinetics of MG-K10 humanized monoclonal antibody in healthy adults

DETAILED DESCRIPTION:
Objectives of the Study

Main objective: To compare the pharmacokinetics of MG-K10 after a single subcutaneous injection in healthy Chinese adult subjects.

Secondary objectives: To evaluate other pharmacokinetic (PK) parameters of MG-K10 after a single subcutaneous injection; The safety and tolerability of a single subcutaneous injection of MG-K10 in healthy Chinese adult subjects were evaluated. To evaluate the immunogenicity of MG-K10 in healthy Chinese adult subjects.

design: The number of cases in this trial was set as 30 cases in test drug (T) group and 30 cases in control drug (R) group, and a total of 60 subjects were enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Participants signed the informed consent form before the study, and fully understood the content, process and possible adverse reactions of the study; Volunteer to participate and be able to complete the study in accordance with the protocol requirements.
2. Chinese healthy adult volunteers, male or female, aged 18-50 years old (inclusive) at the time of signing the informed consent form;
3. During the screening period, the body weight of male volunteers was ≥50 kg; Body weight of women ≥45 kg, and body weight of men and women must not exceed 80 kg (including 80 kg); Body mass index (BMI) in the range of 19.0-26.0kg/m2 (including the boundary value;
4. From the date of signing the informed consent to 6 months after the end of the trial, the volunteers (including male volunteers) had no plans to have children and voluntarily took effective non-drug contraceptive measures, and had no plans to donate sperm or eggs.

Exclusion Criteria:

1. Have any clinically serious disease history or are currently suffering from related diseases, including but not limited to diseases of the digestive system, cardiovascular system, respiratory system (such as asthma, etc.), urinary system, musculoskeletal system, endocrine system, neuropsychiatric system, blood system, immune system and other systems; Have any disorders such as coagulopathy (e.g. hemophilia) or a history of haemorrhagic diseases such as hemorrhoids, acute gastritis or gastric and duodenal ulcers; Patients with severe ocular diseases or acute ocular inflammation (conjunctivitis, blepharitis, keratitis, etc.), dry eye or pruritus; Have herpes virus infection;
2. Those who have participated in and used the trial drug;
3. Lactating and pregnant women, or women of childbearing age volunteers with positive blood pregnancy test;
4. Had a history of dizzy with needles and blood; Or patients with orthostatic hypotension；
5. Patients who had used immunosuppressant or immunopotentiator within 3 months before drug administration;
6. There are birthmarks, scars, tattoos, open wounds at the administration site (around the umbilical cord);

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic: the maximum concentration (Cmax) | 57 days
  Concentration and exposure
Pharmacokinetic: area under the curve of o~t | 57 days
  Concentration and exposure
Pharmacokinetic: area under the curve of o~∞ | 57 days
  Concentration and exposure

SECONDARY OUTCOMES:
Safety evaluation index | 57 days
  Any adverse medical events that occur during a clinical study

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, doctor, Study Director — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China